CLINICAL TRIAL: NCT01038531
Title: Biomarkers of Lung Injury With Low Tidal Volume Ventilation Compared With Airway Pressure Release Ventilation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Allan J. Walkey, Assistant Professor of Medicine, Boston Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H-28944
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Acute Lung Injury; Adult Respiratory Distress Syndrome
Keywords: Acute lung injury (ALI); Adult respiratory distress syndrome (ARDS); Low-tidal-volume strategy; ARDS Net; airway pressure release ventilation (APRV); biomarkers of lung injury
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low-tidal-volume ventilation (Active Comparator): Goal tidal volume is 6 cc/kg ideal body weight.
  Interventions: Other: low-tidal-volume ventilation
- APRV (Experimental): APRV allows spontaneous breathing.
  Interventions: Other: APRV

INTERVENTIONS:
Other: low-tidal-volume ventilation — goal tidal volume of 6 cc/kg ideal body weight
  Arms: low-tidal-volume ventilation
Other: APRV — APRV is a time cycled, inverse-ratio, pressure controlled strategy that allows spontaneous breathing through the respiratory cycle.
  Arms: APRV

SUMMARY:
Acute lung injury (ALI) and the acute respiratory distress syndrome (ARDS) represent a spectrum of clinical syndromes of rapid respiratory system deterioration that are associated with both pulmonary and systemic illness. These syndromes are associated with 30-40% mortality with our current standard of care and are responsible for approximately 75,000 deaths in the US yearly. Current evidence-based care of ALI consists of a strategy of mechanical ventilation utilizing low lung volumes (ARDSNet ventilation) intended to limit further stretch-induced lung injury exacerbated by the ventilator. However, this strategy has been shown to be associated with increased lung injury in a subset of patients and still is associated with about a 30% mortality rate. Airway pressure release ventilation (APRV) is a different, non-experimental strategy of mechanical ventilation currently in routine clinical use. APRV is a pressure-cycled ventilator mode that allows a patient a greater degree of autonomy in controlling his or her breathing pattern than ARDSNet ventilation. Use of APRV has been associated with better oxygenation, less sedative usage, and less ventilator-associated pneumonia in small studies compared with other ventilator modes. However, debate exists over whether APRV might result in decreased or increased ventilator-associated lung injury when compared with ARDSNet ventilation. We intend to implement a randomized, cross over study looking at biomarkers of lung injury in patients with acute lung injury during ventilation with APRV and using the ARDSNet protocol. Our hypothesis is that airway pressure release ventilation is associated with lower levels of lung injury biomarkers than ARDSNet ventilation.

DETAILED DESCRIPTION:
Acute lung injury (ALI) and the acute respiratory distress syndrome (ARDS) represent a spectrum of clinical syndromes of rapid respiratory system deterioration that are associated with both pulmonary and systemic illness. These syndromes are associated with 30-40% mortality with our current standard of care and are responsible for approximately 75,000 deaths in the US yearly. The current evidence-based care consists of a strategy of mechanical ventilation utilizing low lung volumes (ARDSNet ventilation) intended to limit further lung injury from overstretch of the lung induced by the ventilator. However, this strategy has been shown to be associated with continued lung injury in some studies and still is associated with about a 30% mortality rate. Airway pressure release ventilation (APRV) is a different, nonexperimental strategy of mechanical ventilation currently in routine clinical use. APRV allows a patient a greater degree of autonomy in controlling his/her breathing while achieving a higher mean airway pressure (at similar plateau pressures) than that typically achieved with ARDSNet. APRV has been associated with less ventilator-associated pneumonia, better oxygenation, and less sedative usage in small studies when compared with other methods of ventilation. However, debate exists over net effects of APRV with regard to ventilator-associated lung injury. Additionally, we recently completed a study showing that APRV was associated with lower ventilator associated pneumonia (VAP) rates, but this benefit did not appear to be mediated by sedation differences. We hypothesized that the VAP benefits might be mediated by greater lung recruitment and possibly less ventilator-induced lung injury with APRV. We propose a randomized, crossover study looking at biomarkers of lung injury in patients with acute lung injury ventilated with APRV and ARDSNet. Our hypothesis is that airway pressure release ventilation is associated with lower levels of lung injury biomarkers than ARDSNet ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Age > or equal to 18.
* On mechanical ventilation using a volume-controlled mode.
* Admitted to Boston Medical Center Surgical, Medical, or Coronary Intensive Care Unit.
* Meets American-European Consensus Criteria for Acute Lung Injury (ALI) or Acute Respiratory Distress Syndrome.
* Required mechanical ventilator for less than 14 days.
* Met ARDS or ALI criteria for less than 7 days prior to enrollment.
* Assent of primary care team

Exclusion Criteria:

* Do not resuscitate order.
* Increased intracranial pressure.
* Pregnancy (urine pregnancy test for all women of child-bearing age).
* Planned transport out of ICU during planned study protocol.
* Coagulopathy (INR>2.0 or PTT >50).
* Severe thrombocytopenia (platelets <20,000).
* History of obstructive lung disease (asthma and/or COPD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-07; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The study will be powered to detect a decrease in plasma IL-6 levels (pg/ml) from ARDSNet to APRV | 6 hours

SECONDARY OUTCOMES:
Changes in dose of sedation medications | 6 hours
Riker score | 6 hours
Lung mechanics | 6 hours
Oxygenation with APRV versus ARDSNet | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: George O'Connor, MD, Principal Investigator — Boston University Medical College
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States